CLINICAL TRIAL: NCT01786278
Title: The Comparison of Value of Brachytherapy and Endoscopic Stenting With SEMS in Palliative Treatment of Dysphagia Resulting From Adenocarcinoma of the Esophago-Gastric Junction
Brief Title: Comparison Study of Brachytherapy and Endoscopic Stenting for Dysphagia in Esophago-Gastric Junction Cancer
Acronym: BRASTEGAC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lublin (Other)
Collaborators: St Johns' Oncology Center in Lublin (Unknown)
Responsible Party: Principal Investigator, Tomasz Skoczylas, MD, PhD, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGC-DYS-0254/281/2011-MUL; MULEK-0254/281/2011 (Other: Medical University of Lublin)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Adenocarcinoma of the Esophago-gastric Junction
Keywords: adenocarcinoma; esophago-gastric junction; dysphagia; brachytherapy; endoscopic stenting
MeSH Terms: conditions — Adenocarcinoma; Deglutition Disorders | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brachytherapy (Experimental): Single dose of 12 Gy generated using a flexible applicator containing Iridium 192 with the range of irradiation of 1cm from the applicator axis. The extent of irradiation will cover the whole length of cancer stricture and 2cm beyond proximal and distal end of the tumor.
  Interventions: Radiation: Brachytherapy
- Endoscopic Stenting (Other): Endoscopic stenting with partially covered selfexpandable metalic stents positioned across the cancer stricture and extending 2cm proximally and 2cm distally to the proximal and distal end of the tumor, respectively
  Interventions: Procedure: Endoscopic stenting

INTERVENTIONS:
Radiation: Brachytherapy — Single dose of 12 Gy generated using a flexible applicator containing Iridium 192 with the range of irradiation of 1cm from the applicator axis. The extent of irradiation will cover the whole length of cancer stricture and 2cm beyond proximal and distal end of the tumor.
  Arms: Brachytherapy
Procedure: Endoscopic stenting — Endoscopic stenting with partially covered selfexpandable metalic stents positioned across the cancer stricture and extending 2cm proximally and 2cm distally to the proximal and distal end of the tumor, respectively
  Arms: Endoscopic Stenting

SUMMARY:
The objective of the study is comparison of the efficacy and safety of palliative therapy with single-dose brachytherapy or selfexpanding metal stents (SEMS) in malignant dysphagia resulting from adenocarcinoma of the esophago-gastric junction.

DETAILED DESCRIPTION:
Over the past two decades it has been observed a clear trend in the increasing incidence of adenocarcinoma of the esophagus and esophago-gastric junction. More than half of these patients already have inoperable disease at presentation. Most of them need palliative treatment to relieve progressive dysphagia. Presently, endoscopic placement of a covered selfexpanding metal stent is the most commonly used method for treatment of malignant dysphagia. Cancer overgrowth and stent migration are the most common complications of endoscopic stenting and they occur more frequently with longer time from stenting. Specific location at esophago-gastric junction at the end point of the propulsive force after swallow may predispose stents for easier migration to the stomach. Additionally, the advances in chemotherapy have resulted in improved median survival of advanced adenocarcinoma ot the stomach and esophago-gastric junction even up to 10-12 months increasing a potential for higher chance for occurrence of stent complications. Brachytherapy has been proved to be a valuable and durable method to treat malignant dysphagia resulting from esophageal and mainly squamous cell cancer. For many years irradiation was not recommended for adenocarcinoma of the esophagus and esophago-gastric junction due to their putative low sensitivity to radiotherapy. Recently external beam radiation has been incorporated to a combined modality therapy regimens also for adenocarcinoma of the esophagus. Thus, brachytherapy could be an attractive and durable method for improving swallowing in adenocarcinoma of the esophago-gastric junction, as well. Single-dose brachytherapy and endoscopic stenting with SEMS in relieving dysphagia resulting from clearly defined adenocarcinoma of the esophago-gastric junction have not been compared yet.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the esophago-gastric junction defined as adenocarcinoma involving lower esophagus and upper stomach with epicenter of the primary tumor between 5cm above and 5cm below the anatomic esophago-gastric junction
* Inoperable cancer - locally advanced irresectible cancer, distant metastasis or patient's condition does not fit to undergo a curative therapy
* Dysphagia score 2-4
* Performance status 60-100
* Signed informed consent

Exclusion Criteria:

* Esophageal squamous cell carcinoma
* Esophageal adenocarcinoma
* Gastric cancer
* Performance status <60
* Instable cardiocirculatory or respiratory disorder
* Concurrent external beam radiation therapy
* Previous anticancer therapy related to current adenocarcinoma of the esophago-gastric junction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-02 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The highest improvement of dysphagia grade | 1 year
Time to the best swallowing improvement | 1 year
Time to recurrent worsening of swallowing | 1 year
The highest improvement of stricture diameter | 1 year

SECONDARY OUTCOMES:
the procedure related morbidity | 1 year
the procedure related mortality | 1 year
The frequency of dysphagia related additional endoscopic interventions | 1 year
Overall survival | 1 year
Quality of life | 1 year

OTHER OUTCOMES:
Cost analysis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Skoczylas, MD, PhD, Principal Investigator — Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin; Krzysztof Zinkiewicz, MD, PhD, Principal Investigator — Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin; Grzegorz Wallner, Professor, Principal Investigator — Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin; Elżbieta Starosławska, MD, PhD, Principal Investigator — St Johns' Oncology Center in Lublin; Dariusz Kieszko, MD, PhD, Principal Investigator — St Johns' Oncology Center in Lublin
Locations (2):
- Poland (2):
  - Second Department of General & Gastrointestinal Surgery & Oncological Surgery of the Alimantary Tract, Medical University of Lublin, Lublin, Lublin Voivodeship
  - St. John's Cancer Center, Lublin, Lublin Voivodeship